CLINICAL TRIAL: NCT01474174
Title: A Pilot Study of Influenza Vaccine Efficacy in Patients With Central Nervous System Tumors
Brief Title: Trivalent Influenza Vaccine in Preventing Flu in Patients With Central Nervous System Tumors
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00018422; NCI-2011-03033 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 98411 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2011-10-21; First posted 2011-11-18 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Central Nervous System Neoplasm
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Influenza Vaccines; FluMist

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Supportive care (vaccine therapy): Patients receive trivalent influenza vaccine IM on day 0.
  Interventions: Biological: trivalent influenza vaccine; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: trivalent influenza vaccine — Given IM
  Other Names: FluMist; Flushield; Fluvirin; Fluzone; Influenza Vaccine
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies trivalent influenza vaccine in preventing flu in patients with central nervous system (CNS) tumors. Flu vaccine may help the body build an effective immune response and help prevent flu in patients who are receiving chemotherapy for CNS tumors

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary objective of this pilot study is to assess the efficacy of influenza vaccination in patients with central nervous system tumors as defined by a four-fold increase in hemagglutinin inhibition (HI) titers from the pre-vaccination baseline.

SECONDARY OBJECTIVES:

I. A secondary objective of this pilot study is to assess the efficacy of influenza vaccination in patients with central nervous system tumors as defined by a serum post-vaccination HI titer of at least 1:40.

II. The secondary objectives of this pilot study include an assessment of the relationship between a variety of clinical factors and seroconversion following influenza vaccination.

III. Subgroup analyses will include an investigation of seroconversion and treatment (actively receiving chemotherapy, radiation therapy or both), disease status (active treatment vs long term followup), and use and dose of glucocorticoids.

TERTIARY OBJECTIVES:

I. An additional area of interest which will be further explored in this pilot study is an assessment of the relationship between serologic markers of immune function and response to vaccination.

OUTLINE:

Patients receive trivalent influenza vaccine intramuscularly (IM) on day 0.

After completion of study treatment, patients are followed up at 14 days, 21 days, and 3 and/or 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a clinical diagnosis of a primary central nervous system tumor
* Patients must be eligible to receive the influenza vaccine
* Patients must be able to provide written informed consent

Exclusion Criteria:

* Patients unable to receive the influenza vaccine due to history of allergy to egg proteins, allergy to influenza vaccine component, acute febrile illness at the time of proposed vaccine administration, history of clinically or virologically confirmed influenza infection in the previous 6 months, contraindication to intramuscular injections, Guillan-Barré syndrome, or other contraindication to the vaccine
* Patients who have received the 2011-2012 annual influenza vaccine prior to being considered for enrollment on this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with primary central nervous system turmors
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of influenza vaccination in patients with central nervous system tumors as defined by a four-fold increase in HI titers from the pre-vaccination baseline | 6 months
  Seroconversion rate will be defined as the percentage of patients with at least a four-fold increase in HI antibodies between baseline and follow up. Seroprotection rate will be defined as the percentage of patients with a serum HI antibody of at least 1:40. The relationship between seroconversion and various clinical variables including therapy status (active vs longterm follow-up), glucorticoid dose and immune function will be measured. Seroconversion and seroprotection rate comparisons will be made to publish normative data for the general population.

SECONDARY OUTCOMES:
Efficacy of influenza vaccination in patients with central nervous system tumors as defined by a serum post-vaccination HI titer of at least 1:40 | 6 months
Relationship between a variety of clinical factors and seroconversion following influenza vaccination | 6 months
Relationship between serologic markers of immune function and response to vaccination | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Lesser, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States